CLINICAL TRIAL: NCT04708613
Title: Prevalence of Brain Health Versus Neurodegeneration in Former Professional Football Players
Brief Title: University of Pittsburgh Brain Health Initiative
Acronym: BHI
Status: Recruiting | Type: Observational
Sponsor: David Okonkwo, MD, PhD (Other)
Collaborators: National Football League Scientific Advisory Board (Unknown); Avid Radiopharmaceuticals, Inc. (Unknown); Harvard University (Other)
Responsible Party: Sponsor-Investigator, David Okonkwo, MD, PhD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: Brain Health Initiative
Record Dates: First submitted 2021-01-05; First posted 2021-01-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Traumatic Brain Injury
Keywords: Brain Health; Football; Contact Sport; Concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion | interventions — Magnetic Resonance Imaging; Physical Examination; Hematologic Tests; (N-methyl-C-11)-2-(4-methylamino-phenyl)-6-hydroxybenzothiazole; 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole; 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Former Professional Football Players: Former professional football players who played in at least 3 professional seasons, with at least 3 games each season.
  Interventions: Diagnostic Test: Cognitive/Neuropsychological Testing; Diagnostic Test: Vestibular/Ocular-Motor Testing; Diagnostic Test: Sleep Evaluation; Diagnostic Test: MRI, High-Resolution; Diagnostic Test: Health & Physical Exam; Diagnostic Test: Physical Function; Diagnostic Test: Blood Testing and Biomarker Analysis; Diagnostic Test: Applanation Tonometry; Diagnostic Test: PET brain imaging; Drug: [C-11]6-OH-BTA-1; Drug: [F-18]AV-1451
- Control Groups: Friends and brothers of the Former Professional Football Player group.
  Interventions: Diagnostic Test: Cognitive/Neuropsychological Testing; Diagnostic Test: Vestibular/Ocular-Motor Testing; Diagnostic Test: Sleep Evaluation; Diagnostic Test: MRI, High-Resolution; Diagnostic Test: Health & Physical Exam; Diagnostic Test: Physical Function; Diagnostic Test: Blood Testing and Biomarker Analysis; Diagnostic Test: Applanation Tonometry; Diagnostic Test: PET brain imaging; Drug: [C-11]6-OH-BTA-1; Drug: [F-18]AV-1451

INTERVENTIONS:
Diagnostic Test: Cognitive/Neuropsychological Testing — Comprehensive testing of cognitive function and brain health.
Diagnostic Test: Vestibular/Ocular-Motor Testing — A series of tests and questionnaires that asses vestibular function, balance, ocular-motor coordination, and reflexes.
Diagnostic Test: Sleep Evaluation — A full assessment of sleep health, including insomnia (duration, frequency, daytime consequences) and other sleep disorders such as obstructive sleep apnea. Overnight sleep study is included.
Diagnostic Test: MRI, High-Resolution — A high-resolution MRI to provide qualitative and quantitative assessments of brain structure.
Diagnostic Test: Health & Physical Exam — Participants will undergo an executive history and physical exam of all body systems.
Diagnostic Test: Physical Function — These assessments will involve a series of tests and questionnaires that focus on physical function.
Diagnostic Test: Blood Testing and Biomarker Analysis — A blood draw will be performed to measure standard clinical labs as part of a full history and physical, as well as additional analysis of biomarkers indicative of brain health.
  An optional lumbar puncture will be performed and CSF samples (20-30 mL) stored in the NCTC Biorepository until shipment to the CLIA-certified laboratory.
  Both CSF and blood samples will be analyzed for t-tau, p-tau, and Aβ42 and stored for future testing,
Diagnostic Test: Applanation Tonometry — Hearth health is evaluated through testing of arterial stiffness and pulse wave reflections using a high fidelity applanation tonometer.
  Other Names: Continuous arterial pressure
Diagnostic Test: PET brain imaging — PET imaging of the brain using tau and amyloid ligands.
Drug: [C-11]6-OH-BTA-1 — PET imaging of the brain using an amyloid ligand.
  Other Names: Pittsburgh Compound B
Drug: [F-18]AV-1451 — PET imaging of the brain using a tau ligand.
  Other Names: [F-18]T807, LY3191748

SUMMARY:
This project will define the prevalence of brain health (i.e., normal cognitive, neuromotor, behavioral function) in living professional football retirees and group-matched controls through a comprehensive assessment of clinical, neuroimaging, and biomarker measures.

ELIGIBILITY:
Inclusion criteria:

Former professional football player/exposed group:

1. Professional football retiree aged 29-59
2. Played a minimum of 3 professional football seasons, with a minimum of 3 games in each season
3. Fluent in English (translations are not available/validated for most neuropsychological tests)

Control/unexposed group:

1. Age 29-59 male
2. High school education or beyond
3. Fluent in English (translations are not available/validated for most neuropsychological tests)

Exclusion criteria:

Control/unexposed group:

1. Played organized football beyond high school
2. History of severe TBI
3. Current unstable cardiovascular disorder

For both groups:

1. Prior history of psychosis (such as schizophrenia), or other major neurological disorder that would interfere with testing, in the opinion of the primary investigator.
2. Contraindication to MR imaging, such as ferrous metal, pacemakers, or concerns about claustrophobia

Ages: 29 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females will not be included in the study population. Participants will be prior professional football players, age 29-59, that are eligible for a pension. Control participants will be group-matched for age and gender and therefore females will not be included in the study population.
Study Population: 1. Professional Football Players:
     There will be 2 cohorts of former professional football players in this group: (a) random sample, and (b) non-random sample.
     1. Random-Sample participants
        Recruitment of random-sample former professional football players will be conducted via collaboration with the Football Players Health Study (FPHS) at Harvard University. Subjects for the Brain Health Initiative (BHI) will include a random sample of enrollees in the FPHS who meet basic eligibility for BHI.
     2. Non-Random participants:
     We will also enroll a non-random cohort of former professional football players that will be comprised of volunteers.
  2. Controls:
  There will be 3 cohorts of unexposed controls in this group: (a) friends of former players, (b) brothers or former players, and (c) general population. Football players will be invited to refer friend(s) and/or brother(s), but it is not required for participation.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rates of Brain Health versus Cognitive Impairment | 1-week
  The diagnosis of cognitive impairment is based on the ADRC National Alzheimer's Coordinating Center (NACC) criteria for mild cognitive impairment. This criteria is adjudicated following a comprehensive neuropsychological exam, and includes: (1) Self- or informant-reported cognitive complaint, (2) Objective cognitive impairment, (3) Preserved independence in functional abilities, and (4) No dementia.

SECONDARY OUTCOMES:
Clinical Syndromes of Neurodegeneration | 1-week
  The determination of trauma-related neurodegeneration will be based on: 1) presence of cognitive deficits, and/or neuromotor manifestations, and/or behavioral/mood-related symptoms; 2) PET scans demonstrating abnormal amyloid and/or tau deposition; 3) quantitative MR evidence of cortical volume loss and/or white matter injury; and 4) elevated CSF tau/Aβ42 ratio.
  These multiple measures will be combined to arrive at a single overall outcome measure. This will be adjudicated at a blinded Diagnostic Consensus Conference comprised of experts from each field.

CONTACTS AND LOCATIONS:
Overall Officials: David O Okonkwo, MD, PhD, Principal Investigator — University of Pittsburgh Department of Neurological Surgery
Locations (1):
- University of Pittsburgh Department of Neurosurgery, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez OL, Jagust WJ, DeKosky ST, Becker JT, Fitzpatrick A, Dulberg C, Breitner J, Lyketsos C, Jones B, Kawas C, Carlson M, Kuller LH. Prevalence and classification of mild cognitive impairment in the Cardiovascular Health Study Cognition Study: part 1. Arch Neurol. 2003 Oct;60(10):1385-9. doi: 10.1001/archneur.60.10.1385. PMID 14568808
- [Background] Petersen RC. Mild cognitive impairment clinical trials. Nat Rev Drug Discov. 2003 Aug;2(8):646-53. doi: 10.1038/nrd1155. No abstract available. PMID 12904814

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT04708613/SAP_000.pdf